CLINICAL TRIAL: NCT07155083
Title: A Descriptive Survey Study on Firearm Safety Practices, Attitudes, and Perceptions
Brief Title: Firearm Safety Survey
Status: Recruiting | Type: Observational
Sponsor: Vanessa Ng (Other)
Responsible Party: Sponsor-Investigator, Vanessa Ng, Pediatric Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00005069
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Firearm Ownership

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents / Caregivers as Firearm Owner: Parents / caregivers of pediatric patients presenting for surgery stating they are firearm owners.
  Interventions: Other: Survey using a questionnaire.
- Parents / Caregivers as Non-Firearm Owner: Parents / caregivers of pediatric patients presenting for surgery stating they are not firearm owners.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — REDCap Survey

SUMMARY:
The primary objective of this study is to characterize firearm ownership, storage, accessibility, and safety practices. We will also assess perceptions, concerns, and education received on gun safety. This information will be collected through structured surveys given to caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of patients presenting to NCH for any surgery or procedure.

Exclusion Criteria:

* Non legal guardians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents or legal guardians of patients presenting to NCH for any surgery or procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Firearm Ownership | From enrollment to end of perioperative time.
  "Yes" or "No" when asked about firearm ownership.
Demographics | From enrollment to end of perioperative time.
  Descriptive data related to demographics as calculated as frequencies and percentages.

SECONDARY OUTCOMES:
Firearm storage | From enrollment to end of perioperative time.
  Questions related to firearm ownership and storage.
Firearm accessibility | From enrollment to end of perioperative time.
  Questions related to firearm accessibility.
Firearm safety practices | From enrollment to end of perioperative time.
  Questions related to firearm safety practices.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No